CLINICAL TRIAL: NCT04179396
Title: A Phase 1b, Open-label, Parallel Arm Study to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of Oral Rucaparib in Combination With Other Anticancer Agents in Patients With Metastatic Castration Resistant Prostate Cancer
Brief Title: Study of Oral Rucaparib With Other Anticancer Agents in Metastatic Castration Resistant Prostate Cancer Patients (RAMP)
Acronym: RAMP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: pharmaand GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO-338-107
Record Dates: First submitted 2019-11-19; First posted 2019-11-27 (Actual); Results first posted 2023-06-28 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Metastatic Castration Resistant Prostate Cancer
Keywords: CRPC; PARP inhibitor; RAMP; homologous recombination; DNA repair; DNA defect; DNA anomaly; mCRPC; enzalutamide; abiraterone; Zytiga; Xtandi; ADT; AR; ARi
MeSH Terms: interventions — rucaparib; enzalutamide; abiraterone; Abiraterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Oral rucaparib and enzalutamide (Experimental)
  Interventions: Drug: Rucaparib; Drug: Enzalutamide
- Arm B: Oral rucaparib and abiraterone (Experimental)
  Interventions: Drug: Rucaparib; Drug: Abiraterone

INTERVENTIONS:
Drug: Rucaparib — Oral rucaparib will be administered twice daily
  Other Names: Rubraca; CO-338
Drug: Enzalutamide — Enzalutamide will be administered once daily.
  Enrollment into Arm A will be prioritized over Arm B until the objectives for Arm A have been achieved.
  Other Names: Xtandi
  Arms: Arm A: Oral rucaparib and enzalutamide
Drug: Abiraterone — Abiraterone will be administered once daily with prednisone
  Other Names: Zytiga
  Arms: Arm B: Oral rucaparib and abiraterone

SUMMARY:
Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of Oral Rucaparib in Combination with Other Anticancer Agents in Patients with Metastatic Castration Resistant Prostate Cancer

ELIGIBILITY:
Inclusion Criteria:

* Have signed an Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved informed consent form prior to any study-specific evaluation
* Be ≥18 yrs of age at the time the informed consent form is signed
* Be either AR-directed therapy-naive or have received 1-2 lines of AR-directed therapy in the castration-resistant setting.
* Adequate organ function
* ECOG 0 or 1
* Have a histologically or cytologically confirmed adenocarcinoma or poorly differentiated carcinoma of the prostate that is metastatic
* Be surgically or medically castrated, with serum testosterone levels of ≤ 50 ng/dL (1.73 nM)
* Have disease progression after initiation of most recent therapy

Exclusion Criteria:

* Active second malignancy, with the exception of curatively treated non melanoma skin cancer, carcinoma in situ, or superficial bladder cancer
* Have received greater than 2 previous lines of chemotherapy for mCRPC
* Prior treatment with any PARP inhibitor
* Symptomatic and/or untreated central nervous system metastases
* Pre-existing duodenal stent and/or any gastrointestinal disorder or defect that would, in the opinion of the investigator, interfere with absorption of study drug
* Spinal cord compression, symptomatic and/or untreated central nervous system (CNS) metastases or leptomeningeal disease. Patients with asymptomatic previously treated CNS metastases are eligible provided they have been clinically stable for at least 4 weeks
* Any clinically significant cardiovascular disease
* Taking any concomitant medications or herbs that could interfere or interact with the study drug

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2023-01-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Piedmont Cancer Institute, P.C., Atlanta, Georgia
  - University of Minnesota, Minneapolis, Minnesota
  - Urology Associates, P.C., Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets for study results will be made available to qualified researchers in compliance with applicable privacy laws and data protection regulations.
  Data will be provided by Clovis Oncology.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available to qualified researchers after the primary, secondary, and/or exploratory outcomes of the study are reported or published and for 1 year thereafter.
Access Criteria: Requests for de-identified datasets will be made available to qualified researchers following submission of a methodologically sound proposal to medinfo@clovisoncology.com.

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Oral Rucaparib and Enzalutamide: Rucaparib: Oral rucaparib will be administered twice daily
  Enzalutamide: Enzalutamide will be administered once daily.
  Enrollment into Arm A will be prioritized over Arm B until the objectives for Arm A have been achieved.
- Arm B: Oral Rucaparib and Abiraterone: Rucaparib: Oral rucaparib will be administered twice daily
  Abiraterone: Abiraterone will be administered once daily with prednisone
  Arm B was never opened
Period: Overall Study
Arm/Group | Arm A: Oral Rucaparib and Enzalutamide | Arm B: Oral Rucaparib and Abiraterone
Started | 8 | 0
Completed | 8 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Arm B was never open to enrollment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Oral Rucaparib and Enzalutamide | Arm B: Oral Rucaparib and Abiraterone | Total
Number analyzed (Participants) | 8 | 0 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 0 | 3
  >=65 years | 5 | 0 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 0 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 0 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the PK of Rucaparib in Combination With Other Anticancer Agents for mCRPC.
Description: Cmin of rucaparib and its metabolite. Rucaparib only run-in Cmin includes run-in D6, D7 and Cycle 1 D1. All of these samples were collected following rucaparib monotherapy. Rucaparib and other anticancer agent Combination Cmin includes Cycle 1 (D8, D15, and D22).
Time Frame: 1 week rucaparib only run-in and 1 cycle (28 days) of combination treatment
Population: Arm B was never open
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Arm A: Oral Rucaparib and Enzalutamide | Arm B: Oral Rucaparib and Abiraterone
Number analyzed (Participants) | 7 | 0
ng/ml
  Cmin of rucaparib during 1-week rucaparib only run-in | 1345 (529) |
  Cmin of rucaparib metabolite M324 during 1-week rucaparib only run-in | 233 (103) |
  Cmin of rucaparib during 1st cycle of rucaparib enzalutamide combo treatment | 1558 (510) |
  Cmin of rucaparib metabolite M324 during 1st cycle of rucaparib enzalutamide combo treatment | 311 (161) |

2. Primary Outcome: Incidence of Dose-Limiting Toxicities (DLTs) in Participants Taking Rucaparib in Combination With Other Anticancer Agents for mCRPC
Description: A DLT is defined according to criteria specified in the protocol and assessed by the investigator, based on toxicity grade (according to the NCI CTCAE v5.0), clinical significance, and possible relationship to the study drug combination. The toxicity cannot be a recognized adverse effect of enzalutamide, abiraterone or prednisone/prednisolone and/or attributable to mCRPC or mCRPC-related processes under investigation.
Time Frame: First 2 cycles of rucaparib combination treatment (56 days) for Arm A
Population: Number of participants deemed DLT-evaluable
  Arm B was never opened
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Oral Rucaparib and Enzalutamide | Arm B: Oral Rucaparib and Abiraterone
Number analyzed (Participants) | 6 | 0
Participants | 0 | 0

3. Secondary Outcome: Preliminary Overall Confirmed Response Rate (ORR) of Rucaparib in Combination With Other Anticancer Agents for mCRPC.
Description: The ORR is defined as the proportion of patients with a documented and confirmed best overall response of complete response (CR) or partial response (PR) per mRECIST v1.1 as assessed by the investigator using local standardized radiological methods e.g. CT, MRI, etc. A complete response (CR) is defined as complete disappearance of all target and non-target lesions together with normalization of tumor biomarkers. A partial response (PR) represents at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum LD with non-progression of non-target lesions and no new lesions. Overall Response (OR) = CR + PR. A confirmed CR or PR is a response that is maintained and documented on a subsequent tumor assessment at least 4 weeks after initial response. PSA response per PCWG3 criteria is a confirmed PSA response (≥ 50% decrease from baseline) as reflected by local laboratory measurements.
Time Frame: 2 years to complete
Population: Preliminary ORR could only be evaluated in patients with measurable target lesions at baseline. Only 1 patient had measurable disease at baseline that could be evaluated for a tumor response.
  Arm B was never opened
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Oral Rucaparib and Enzalutamide | Arm B: Oral Rucaparib and Abiraterone
Number analyzed (Participants) | 8 | 0
Participants
  Patients with measurable disease at baseline and a confirmed response of CR or PR by RECISTv1.1 | 1 | 0
  Patients inevaluable for response by RECISTv1.1 | 7 | 0

ADVERSE EVENTS:
Time Frame: 2 years, 5 months
Description: Adverse events collected from first dose of any study drug to 28 days after last dose of study drug, or data cut date where that is earlier. If a patient experienced the same preferred term multiple times, then the patient was counted only once for that preferred term. Arm B was never opened to enrollment
Arm/Group | Arm A: Oral Rucaparib and Enzalutamide | Arm B: Oral Rucaparib and Abiraterone
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/8 | 0/0
Other Adverse Events (participants affected / at risk) | 8/8 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Oral Rucaparib and Enzalutamide (N=8) | Arm B: Oral Rucaparib and Abiraterone (N=0)
Contrast media reaction (Immune system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Oral Rucaparib and Enzalutamide (N=8) | Arm B: Oral Rucaparib and Abiraterone (N=0)
Anaemia (Blood and lymphatic system disorders) | 5 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 0
Eructation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 7 | 0
Retching (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Fatigue (General disorders) | 7 | 0
Feeling abnormal (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Contrast media allergy (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 0
Blood creatinine increased (Investigations) | 2 | 0
Blood urea increased (Investigations) | 1 | 0
Creatinine renal clearance decreased (Investigations) | 2 | 0
Lymphocyte count decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 2 | 0
Platelet count decreased (Investigations) | 4 | 0
Protein total decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 2 | 0
White blood cell count decreased (Investigations) | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 6 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 2 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 5 | 0
Syncope (Nervous system disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Enrollment in the trial was terminated early however sufficient PK and safety data were collected to complete the key objective of elucidating the potential for drug-drug interaction by evaluating PK as well as safety and tolerability of the rucaparib/enzalutamide combination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor's agreements with investigators require proposed public disclosures of trial results to be submitted to Sponsor for review prior to publication. Sponsor may request deletion of confidential information or a delay in publication to address intellectual property concerns, but Sponsor may not suppress publication of the trial results indefinitely. Sponsor may request delay of a single-center publication until after the release of a multi-site publication or an agreed upon period of time.

DOCUMENTS (2):
  • Study Protocol (2022-01-19): https://cdn.clinicaltrials.gov/large-docs/96/NCT04179396/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-02): https://cdn.clinicaltrials.gov/large-docs/96/NCT04179396/SAP_001.pdf